CLINICAL TRIAL: NCT05650970
Title: "Investigation of the Effect of Radial Nerve Mobilization on Pain, Function and Grip Strength in Patients With Hand Thumb Osteoarthritis"
Brief Title: Radial Nerve Mobilization in Hand Thumb Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Sedanur Güngör, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1117
Record Dates: First submitted 2022-11-28; First posted 2022-12-14 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis Thumb; Joint Diseases; Radial Neuropathy
Keywords: osteoarthritis; mobilization; radial nerve; carpometacarpal joint; thumb
MeSH Terms: conditions — Joint Diseases; Radial Neuropathy; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: The 40 people included in the study will be equally placed in the control and study groups in the order they applied to the clinic. Individuals in the two study groups will be included in an exercise program two days a week, accompanied by a physiotherapist for 4 weeks. The only difference between the groups is the content of the treatment programs.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routinely treated control group (Active Comparator): Unlike the study group, radial nerve mobilization will not be included in the treatment program of this group. only massage, ice and activity modification training will be included.
  Interventions: Other: routine therapy
- radial nerve mobilization study group (Experimental): The treatment program of this group will include massage, radial nerve mobilization, ice and activity modification training.
  Interventions: Other: radial nerve mobilization exercise

INTERVENTIONS:
Other: routine therapy — Routine treatment program including massage, ice and activity training applied to hand thumb osteoarthritis patients
  Arms: routinely treated control group
Other: radial nerve mobilization exercise — Radial nerve mobilization exercise in addition to the routine treatment program applied to patients with hand thumb osteoarthritis
  Arms: radial nerve mobilization study group

SUMMARY:
Hand-thumb carpometacarpal (1st CMC) joint osteoarthritis is defined as the degeneration occurring between the articular surfaces of the 1st metacarpal bone and the trapezium bone. This degeneration causes deterioration in the cartilage tissue that forms the joint structure, and as a result, patients primarily complain of pain and related loss of function. Clinical observations and studies have shown that the level of pain expressed by patients is not always compatible with the amount of degeneration in the joint. In addition, it has been clearly stated in the studies that the pain complaints of the patients are not only due to the changes in the joint, but the irritation of the nerves that receive the sensation of this joint is also effective in the level of pain. In line with the findings of the studies on this subject, mobilization exercise for the relevant nerve is included in the treatment programs of patients diagnosed with 1st CMC joint osteoarthritis in the clinic for a while. The investigators observed that the radial nerve mobilization exercise given during the process contributed to the improvement in the pain level of the patients. The investigators planned our study because there was no publication in the literature examining this effect. This study aims to investigate the effect of radial nerve mobilization exercise on pain level, functional status, and grip strength of patients diagnosed with 1st CMC joint osteoarthritis.

DETAILED DESCRIPTION:
Patients will be included in the study voluntarily, they will be informed about the study before their evaluation, and their consent to participate in the study will be obtained with an informed consent form. Evaluations will begin after patient consent is obtained. The patient's age, gender, height, body weight, dominant side, symptomatic side, surgical history, previous treatments for the disease, and the duration of pain will be recorded. Physical assessments will then follow. Evaluations will be made twice, before treatment and at the end of 4 weeks of treatment.

The pain level, coarse and fine grip strength, fine dexterity, functional status, and disability level of the patients will be evaluated. The evaluations made will be the same for the study and control groups. The pain level of the participants will be questioned with the visual analog scale (VAS) in three situations: rest, activity, and night, and will be recorded in cm. Factors that increase and decrease pain will also be questioned and recorded.

Coarse grip strength will be evaluated with a hydraulic hand dynamometer (Jamar®) and fine grip strength will be evaluated with a pinch meter. Grip strength measurement will be made in the standard sitting position determined by the American Association of Hand Therapists. This is the position in which the participant holds the evaluated arm next to the torso, with the elbow flexed to 90 degrees and the wrist in a neutral position. It has been shown in studies that the position of this test has high reliability for the results. During the assessment, the patient will sit in a supported chair. Fine grip strength will be measured in bipod pinch and lateral grip positions. The grip strength measurements will be repeated 3 times in a row for both sides and the patient will be asked to squeeze as hard as possible. The average value of the measurement results will be taken and recorded in kilograms.

The 9-Hole Peg test will be used to evaluate the functional status and fine dexterity of the hand. During this evaluation, the patient will sit in a comfortable position. Both parties will be evaluated separately. The patient will be taught the test to be performed first and will be allowed to make a trial. He will be asked to quickly reinsert all the sticks, starting from the position inserted in the holes and removing the last one as fast as he can using only the first two fingers of the side being evaluated. The total removal and insertion time will be recorded in seconds for each side separately.

The FIHOA (Functional Index of Hand Osteoarthritis) questionnaire will be used to evaluate the level of disability specific to the disease. The questionnaire consists of 10 items containing statements about hand use in daily life, and each item is scored between 0-3 points (0: no difficulty, 1: mild difficulty, 2: quite difficult, 3: impossible) according to the difficulty level. Total score 0-30 points. varies between As a result of this survey, a low score represents a better function, while a high score represents a worse function. It has been shown in studies that it has a high correlation with other osteoarthritis-specific questionnaires, and its validity and reliability. The Turkish version was found to be valid and reliable by Kılıçoğlu et al.

The Michigan Hand Outcomes Questionnaire (MHQ) is a questionnaire used in the general evaluation of the use of the hand on both sides and right-left separately in daily life. In addition, the MHQ has been shown to have good reliability, validity, and responsiveness in patients with 1st CMC joint osteoarthritis. Its use in this patient population is recommended as an appropriate assessment tool. The questionnaire evaluates pain, function, aesthetic appearance, and satisfaction as sub-parameters. Since the MHQ measures function/satisfaction, the higher the score, the higher the functionality/satisfaction a person reports. The validity of the Turkish version of the questionnaire was demonstrated by Öksüz et al. Patients in both groups will be included in the treatment program in the clinic for 4 weeks, 2 sessions per week. On the days when the patients do not come to the clinic, the treatment will continue as a home program. Patients will be asked to do the same treatment program as in the clinic, 3 times a day at home. Different from the control group, nerve mobilization exercises will also be included in the treatment program of the study group. All other practices and training will be done by the same physiotherapist for both groups. Nerve mobilization is a treatment consisting of stretching and sliding techniques that is frequently used in the clinic. The sliding technique is one of the neurodynamic techniques and unlike the stretching technique, it does not cause a decrease in the fluid flow and blood circulation in the nerve. Within the scope of our study, nerve mobilization exercise to be applied to patients with 1st CMC joint osteoarthritis is routinely used in the clinic as a part of conservative treatment. It has been observed that exercises for the nerve innervating the 1st CMC joint have a positive effect on the pain level of the patients in the clinic. Based on this situation, the effect of exercises on the improvement of pain level, function, and strength in patients will be investigated. The content of the treatment program given to the groups consists of the following:

* Patient education: During the treatment, patients will be told not to use their hands in heavy work and not to do any other practice other than treatment. It will be examined how the patients use their hands during the day in line with their daily life activities, hobbies, and profession, and the correct grip positions will be taught. Activity modification will be made (if necessary) for the use of the hand in the workplace.
* Activity modification and teaching correct grip/grip techniques: Patients will be taught correct holding techniques with objects of different sizes and shapes and will be instructed to maintain this position during their daily activities. By questioning their activities, hobbies, and occupation, modifications will be suggested for situations that will exacerbate the pain.
* Classical massage: It will be applied on the line where the superficial branch of the radial nerve passes in the forearm, including only the thumb. It will be done to provide relaxation in the tissue, to reduce pain with mechanical stimulation, to reduce edema that develops due to degeneration around the nerve and joint, and accordingly to contribute to healing.
* Nerve mobilization exercise: Radial nerve mobilization can be performed in two ways: from the isolated wrist (ulnar-radial deviation in the form of a fist by grasping the thumb in the palm) and in combination with the wrist-elbow (starting in the anatomical stance position, while the elbow is in extension, the wrist is in ulnar deviation, while the elbow is in flexion, the wrist is in radial deviation). will be done. This exercise will only be included in the study group.
* Ice application: At the end of the treatment, ice will be applied to the sensory area of the superficial branch of the radial nerve for 10-12 minutes. During the treatment, patients will be told not to use their hands in heavy work and not to do any other application other than treatment.

At the end of the study, if the nerve mobilization exercise shows a significant curative effect on the patients, the patients in the control group will also be given nerve mobilization exercises in the presence of a physiotherapist twice a week for 4 weeks, and they will be asked to do the same exercises 3 times a day within the home programs on the other days.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Hand-thumb Osteoarthritis Disease Must have pain

Exclusion Criteria:

Wrist surgery history Poor communication Poor mental state

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Pain level assessment at rest, activity and at night with a visual analog scale (VAS) | 4 week
  Patients will be asked to mark the value corresponding to the pain levels they feel in three different situations, resting, activity and night, on a line drawn with a length of 10 cm. The level of the marked point will be recorded in cm. 0 point corresponding to the lowest value will be described as I have no pain, 10 points corresponding to the highest value will be described as I have extreme unbearable pain.

SECONDARY OUTCOMES:
gross and fine grip strength assessment | 4 week
  Grip strength will be measured with Jamar® brand hydraulic hand dynamometer and fine grip strength will be measured with Baseline brand pinch gauge. During the grip strength measurement, the evaluated arm of the participant is at the side of the trunk, the elbow is in 90 degrees flexion, the forearm is in the pronation-supination position, and the wrist is in the neutral position. During the measurement, the patient sits in a supported chair with the knees flexed to 90° and the feet in full contact with the floor. The same command will be given to all patients during the measurement. Patients will be asked to squeeze the dynamometer with full force three times in a row. It will be recorded in kilograms (kg) by averaging the three measurements. Measurements will be made bilaterally in all patients.
Functional status assessment with FIHOA (Functional Index of Hand Osteoarthritis) and (Michigan Hand Outcomes Questionnaires-MHOQ) | 4 week
  The FIHOA questionnaire will be used to assess the level of disability specific to the disease. It consists of 10 items containing statements about the use of hands in daily life. Each item is scored between 0-3 points according to skill level (0: no difficulty, 1: mild difficulty, 2: quite difficult, 3: impossible). The total score varies between 0-30 points. As a result of this survey, a low score represents a better function, and a high score represents a worse function.
  The MHOQ is a questionnaire used to evaluate the general use of the hand in daily life. At the beginning of the questionnaire, patients will be asked to answer the statements considering their general condition in the last week. The questionnaire consists of sub-parameters that question pain, function, work, aesthetic appearance, and satisfaction separately. Because the MHOQ measures function/satisfaction, the higher the score on the survey result, the higher the individual's reported functioning/satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Health Science Faculty Physiotherapy and Rehabilitation Department, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sousa-Santos AR, Amaral TF. Differences in handgrip strength protocols to identify sarcopenia and frailty - a systematic review. BMC Geriatr. 2017 Oct 16;17(1):238. doi: 10.1186/s12877-017-0625-y. PMID 29037155
- [Background] Bohannon RW, Bubela DJ, Magasi SR, Gershon RC. Relative reliability of three objective tests of limb muscle strength. Isokinet Exerc Sci. 2011;19(2):10.3233/IES-2011-0400. doi: 10.3233/IES-2011-0400. PMID 24339479
- [Background] Poole JL. Measures of hand function: Arthritis Hand Function Test (AHFT), Australian Canadian Osteoarthritis Hand Index (AUSCAN), Cochin Hand Function Scale, Functional Index for Hand Osteoarthritis (FIHOA), Grip Ability Test (GAT), Jebsen Hand Function Test (JHFT), and Michigan Hand Outcomes Questionnaire (MHQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S189-99. doi: 10.1002/acr.20631. No abstract available. PMID 22588744
- [Background] Dreiser RL, Maheu E, Guillou GB, Caspard H, Grouin JM. Validation of an algofunctional index for osteoarthritis of the hand. Rev Rhum Engl Ed. 1995 Jun;62(6 Suppl 1):43S-53S. PMID 7583182
- [Background] Moe RH, Garratt A, Slatkowsky-Christensen B, Maheu E, Mowinckel P, Kvien TK, Kjeken I, Hagen KB, Uhlig T. Concurrent evaluation of data quality, reliability and validity of the Australian/Canadian Osteoarthritis Hand Index and the Functional Index for Hand Osteoarthritis. Rheumatology (Oxford). 2010 Dec;49(12):2327-36. doi: 10.1093/rheumatology/keq219. Epub 2010 Aug 11. PMID 20702486

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT05650970/Prot_SAP_000.pdf